CLINICAL TRIAL: NCT00366028
Title: Strengthening Organization to Implement Evidence-based Clinical Practice
Brief Title: Increasing Evidence-based Clinical Practices in VA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Factorial | Masking: None
Other Study IDs: IMV 04-055
Record Dates: First submitted 2006-08-16; First posted 2006-08-18 (Estimated); Results first posted 2014-09-26 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2014-05

CONDITIONS: Hand Washing
Keywords: Organization Innovation; Diffusion of Innovation; Evidence-based Medicine; Infection Control

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Organizational Model (Other): Organizational Model: Participants in this arm of the study will receive information regarding the organizational model and work closely with the research team throughout the project to implement various aspects of the model. Participants in this arm of the study will be interviewed and participate in the data feedback portion of the study as well.
  Interventions: Behavioral: Organization Model; Behavioral: Data Feedback Model
- Data Feedback (Other): Data Feedback Only: Participants in this arm will be interviewed periodically and participate in the data feedback portion of the study.
  Interventions: Behavioral: Data Feedback Model

INTERVENTIONS:
Behavioral: Organization Model — The organizational model contains three components: leadership support, a multidisciplinary redesign team, and management structures and processes to link the two.
  Arms: Organizational Model
Behavioral: Data Feedback Model — The research team will periodically interview the facilities and provide them with reported hand hygiene data.

SUMMARY:
Evidence-based clinical practices (EBCPs) are often not widely adopted, despite extensive efforts to influence individual practitioners to use them. The aim of the project is to work with Veterans Integrated Service Networks (VISN) 1, 10, and 23 and their medical centers to create and test organizations that facilitate the use of EBCPs. The research objectives are to: Test the effectiveness of the proposed organizational model in comparison with a more limited data-feedback strategy in improving system use of a selected EBCP; Identify and analyze organizational factors that affect model implementation; Test the feasibility of intervention activities to introduce and support the model.

DETAILED DESCRIPTION:
Background:

The Veterans Health Administration (VHA) needs to develop efficient ways to broadly implement evidence based practices and foster a learning organization culture that systematically and continuously applies research to improve VA healthcare. Recognizing this need, VHA Health Services Research and Development (HSR&D) invited applications in the fall of 2003 for collaboration HSR&D investigators and Integrated Service Networks (VISNs) on a) implementing and evaluating an evidenced-based interventions or b) undergoing and evaluating an organizational or structural change to transform the VISN in to a learning organization that can efficiently implement evidence-based practices. Collaborations are intended to help improve clinical services locally within participating VISNs and provide templates for expanding successful changes nationwide.

Objectives:

Despite recognition that successful implementation of evidence-based clinical practices (EBCPs) usually depends on the on the structure and processes of the larger healthcare organization in which new clinical practices are introduced, the processes and dynamics of implementation are not well understood. The aim of this project was to deepen that understanding by testing an organizational model that we hypothesized would strengthen the ability of healthcare organizations to implement evidence-based clinical practices. The research objectives were to: - Test the hypothesis that medical centers with high fidelity to the organizational model would be more successful in improving system use of a selected EBCP; - Identify and analyze organizational factors that affect model implementation; - Test the feasibility of intervention activities to introduce and support the model.

Methods:

The three-year study used a mixed-methods pre-post comparison-group design to implement and evaluate the organizational model in medical centers in 3 VISNs in the Department of Veterans Affairs. The model posits that the implementation of evidence-based practices will be enhanced through the presence of three interacting components in the organization: 1) active leadership commitment to quality, 2) robust clinical process redesign to incorporate evidence-based practices into routine operations, and 3) use of management structures and processes to support and align redesign. The target clinical practice was hand-hygiene compliance. One VISN was randomly assigned to the intervention arm that implemented the organizational model; two VISNs were assigned to a comparison arm that participated in a more limited data feedback strategy. Measures included: 1) ratings of implementation fidelity, as measured on a 0-4 scale at the site level supported by narrative evidence by research team; 2) percent compliance with national hand-hygiene guidelines for each site, as measured through structured observations by medical center staff; 3) staff ratings of team effectiveness and facility emphasis on quality, as measured through a written survey; and 4) factors affecting model implementation, as identified qualitatively through interviews and quantitatively through staff surveys

Status:

Data collection and analysis is complete. Manuscript preparation is ongoing.

ELIGIBILITY:
Inclusion Criteria:

VA employees of VISNs 1, 10 and 23 working in participating clinical units or holding a leadership position in medical centers identified by facility leadership for participation in the study.

Exclusion Criteria:

Must have operational proficiency in English. All to be interviewed and surveyed will hold professional positions in VA, so this is not expected to be a major barrier to inclusion.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1624 (Actual)
Dates: Start 2006-01; Primary Completion 2008-08 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol VanDeusen-Lukas, EdD, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (1):
- VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts, United States

REFERENCES:
- [Result] VanDeusen Lukas C, Engle RL, Holmes SK, Parker VA, Petzel RA, Nealon Seibert M, Shwartz M, Sullivan JL. Strengthening organizations to implement evidence-based clinical practices. Health Care Manage Rev. 2010 Jul-Sep;35(3):235-45. doi: 10.1097/HMR.0b013e3181dde6a5. PMID 20551771

RESULTS

PARTICIPANT FLOW:
Groups:
- Organizational Model: This arm is considered the intervention arm. Participants in this arm of the study will receive information regarding the organizational model and work closely with the research team throughout the project to implement various aspects of the model.
  Organization Model: The organizational model contains three components: leadership support, a multidisciplinary redesign team, and management structures and processes to link the two.
- Data Feedback: This arm is considered the control arm. Participants in this arm will be interviewed periodically and participate in the data feedback portion of the study but will not undergo any active intervention pertaining to the organizational model.
  Data Feedback Model: This is considered the non-intervention arm. The research team will periodically interview the facilities and provide them with reported hand hygiene data.
Period: Overall Study
Arm/Group | Organizational Model | Data Feedback
Started | 889 | 735
Completed | 889 | 735
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Organizational Model: Participants in this arm of the study will receive information regarding the organizational model and work closely with the research team throughout the project to implement various aspects of the model.
  Organization Model: The organizational model contains three components: leadership support, a multidisciplinary redesign team, and management structures and processes to link the two. The research team will periodically interview the facilities and provide them with reported hand hygiene data.
- Data Feedback: Participants in this arm will be interviewed periodically and participate in the data feedback portion of the study but will not undergo any active intervention pertaining to the organizational model.
  Data Feedback Only Model: The research team will periodically interview the facilities and provide them with reported hand hygiene data.
- Total: Total of all reporting groups
Arm/Group | Organizational Model | Data Feedback | Total
Number analyzed (Participants) | 889 | 735 | 1624
Age, Categorical [Count of Participants; unit: Participants] — Age was not collected as it was not pertinent to the outcome of the study.
  Participants
    <=18 years | NA — Age was not collected as it was not pertinent to the outcome of the study. | NA — Age was not collected as it was not pertinent to the outcome of the study. | NA — Total not calculated because data are not available (NA) in one or more arms.
    Between 18 and 65 years | NA — Age was not collected as it was not pertinent to the outcome of the study. | NA — Age was not collected as it was not pertinent to the outcome of the study. | NA — Total not calculated because data are not available (NA) in one or more arms.
    >=65 years | NA — Age was not collected as it was not pertinent to the outcome of the study. | NA — Age was not collected as it was not pertinent to the outcome of the study. | NA — Total not calculated because data are not available (NA) in one or more arms.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — Gender was not collected as it was not pertinent to the outcome of the study. | NA — Gender was not collected as it was not pertinent to the outcome of the study. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male | NA — Gender was not collected as it was not pertinent to the outcome of the study. | NA — Gender was not collected as it was not pertinent to the outcome of the study. | NA — Total not calculated because data are not available (NA) in one or more arms.

OUTCOME MEASURES:

1. Primary Outcome: Fidelity to the Organizational Model
Description: Final fidelity to the Organizational Model was assessed by averaging scores for each component of the model. Scores ranged from 0 (no evidence of that factor present) to 4 (factor fully present and used as intended). The 3 main components of the model included 1) active leadership commitment to quality, 2) robust clinical process redesign to incorporate evidence-based practices into routine operations, and 3) use of management structures and processes to support and align redesign. Scores for each component of the model were measured by the study team using structured rating instruments based on data collected during interviews.
  Sites with an overall fidelity score above 3.0 were considered to have high fidelity to the organizational model.
Time Frame: Fidelity was assessed at the end of the 3 year study.
Population: This outcome measure was only assessed at the site (facility) level.
Measure: Number; unit: units on a scale
Units Other Than Participants: Facilities
Groups:
- Organizational Model: Participants in this arm of the study received information regarding the organizational model and worked closely with the research team throughout the project to implement various aspects of the model.
  Organization Model: The organizational model contains three components: leadership support, a multidisciplinary redesign team, and management structures and processes to link the two.
  The Intervention Arm included 889 individual participants across 7 study sites (medical centers).
- Data Feedback: Participants in this arm were interviewed periodically and participated in the data feedback portion of the study but did not undergo any active intervention pertaining to the organizational model.
  Data Feedback Model: This is considered the non-intervention arm. The research team periodically interviewed the facilities and provided them with reported hand hygiene data.
  The Control Arm included 735 individual participants across 9 study sites (medical centers) in total. Only 5 of the study sites are included in the reporting of outcome data due to incomplete data at 4 of the study sites.
Arm/Group | Organizational Model | Data Feedback
Number analyzed (Participants) | 889 | 735
Number analyzed (Facilities) | 7 | 5
units on a scale
  Site A | 3.95 | NA — This site is not in the Organizational Model Arm.
  Site B | 3.38 | NA — This site is not in the Organizational Model Arm.
  Site C | 3.23 | NA — This site is not in the Organizational Model Arm.
  Site D | 3.17 | NA — This site is not in the Organizational Model Arm.
  Site E | 2.15 | NA — This site is not in the Organizational Model Arm.
  Site F | 1.98 | NA — This site is not in the Organizational Model Arm.
  Site G | 1.42 | NA — This site is not in the Organizational Model Arm.
  Site H | NA — This site is not in the Data Feedback Arm. | 2.30
  Site I | NA — This site is not in the Data Feedback Arm. | 1.62
  Site J | NA — This site is not in the Data Feedback Arm. | 1.52
  Site K | NA — This site is not in the Data Feedback Arm. | 1.40
  Site L | NA — This site is not in the Data Feedback Arm. | 1.30

2. Primary Outcome: Effect Size of Improvement in Hand Hygiene Compliance
Description: The effect size of improvement in hand-hygiene compliance was calculated by comparing the baseline three-month periods to the last three-month periods of the study. To evaluate the statistical significance of changes in proportion adherence over time, we ran a weighted least squares regression model with time (i.e. month) as the independent variable and adherence proportion as the dependent variable. The sample size in each data collection period was used as the weight. Our interest is in the statistical significance of the coefficient associated with time. To evaluate the practical significance of the change pre and post intervention, we examined the effect size associated with the change in proportion adherence in the first 3-month period of data collection and the last 3-month period. Effect size was calculated as 2*arcsin(sqr(p2)) - 2*arcsin(sqr(p1)). Using Cohen's criteria, an effect size of .2 is interpreted as small, .5 as medium and .8 as large.
Time Frame: 3 months pre and post study intervention
Population: This outcome measure was only assessed at the site (facility) level.
Measure: Number; unit: effect size
Units Other Than Participants: Facilities
Groups:
- Organizational Model: Participants in this arm of the study received information regarding the organizational model and worked closely with the research team throughout the project to implement various aspects of the model.
  Organization Model: The organizational model contains three components: leadership support, a multidisciplinary redesign team, and management structures and processes to link the two.
  The Intervention Arm included 7 study sites (medical centers). Of the 7 sites there were 4 with high fidelity to the Organizational Model and 3 with low fidelity to the Organizational Model.
- Data Feedback: Participants in this arm were interviewed periodically and participated in the data feedback portion of the study but did not undergo any active intervention pertaining to the organizational model.
  Data Feedback Model: This is considered the non-intervention arm. The research team periodically interviewed the facilities and provided them with reported hand hygiene data.
  The Control Arm included 9 study sites (medical centers) in total. Only 5 of the study sites are included in analysis of this outcome measure due to incomplete hand hygiene data at 4 of the study sites. Of the 5 study sites included, there were 2 sites with high fidelity to the Organization Model and 3 sites with low fidelity to the Organizational model, even though the model was not specifically introduced to the control arm.
Arm/Group | Organizational Model | Data Feedback
Number analyzed (Participants) | 7 | 5
Number analyzed (Facilities) | 7 | 5
effect size
  Site A | 0.67 | NA — This site was not in the Organizational Model Arm.
  Site B | 0.48 | NA — This site was not in the Organizational Model Arm.
  Site C | 0.92 | NA — This site was not in the Organizational Model Arm.
  Site D | 0.52 | NA — This site was not in the Organizational Model Arm.
  Site E | 0.14 | NA — This site was not in the Organizational Model Arm.
  Site F | 0.14 | NA — This site was not in the Organizational Model Arm.
  Site G | -0.22 | NA — This site was not in the Organizational Model Arm.
  Site H | NA — This site was not in the Data Feedback Arm. | 0.77
  Site I | NA — This site was not in the Data Feedback Arm. | 0.61
  Site J | NA — This site was not in the Data Feedback Arm. | -0.26
  Site K | NA — This site was not in the Data Feedback Arm. | 0.05
  Site L | NA — This site was not in the Data Feedback Arm. | 0.24

ADVERSE EVENTS:
Description: No adverse events were collected.
Groups:
- Organizational Model: This arm is considered the intervention arm. Participants in this arm of the study will receive information regarding the organizational model and work closely with the research team throughout the project to implement various aspects of the model.
  Organization Model: The organizational model contains three components: leadership support, a multidisciplinary redesign team, and management structures and processes to link the two.
  Data Feedback Model: This is considered the non-intervention arm. The research team will periodically interview the facilities and provide them with reported hand hygiene data.
Arm/Group | Organizational Model | Data Feedback
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes